CLINICAL TRIAL: NCT04700930
Title: CBD Cigarettes Instead of Normal Cigarettes Against Enforcement Measures, for Improved Acute Treatment and for Harm Reduction of Smoking - Innovative Treatment for Schizophrenia
Brief Title: CBD Cigarettes Instead of Normal Cigarettes as Innovative Treatment for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Principal Investigator, Prof. Stefan Borgwardt, Principle Investigator, Clinical Professor, Prof. Dr. med., Psychiatric Hospital of the University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01111
Record Dates: First submitted 2020-09-21; First posted 2021-01-08 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia and Other Psychotic Disorders; Harm Reduction
MeSH Terms: conditions — Schizophrenia; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD (Experimental): Patients receive CBD cigarettes additionally to standard psychiatric care including neuroleptic medication
  Interventions: Other: CBD-Cigarettes
- Non-CBD (No Intervention): Patients recieve standard psychiatric care including neuroleptic medication

INTERVENTIONS:
Other: CBD-Cigarettes — CBD-Cigarettes instead of normal Cigarettes: The participants in this arm receive CBD-Cigarettes which are then inhaled/smoked instead of their normal tobacco cigarettes
  Arms: CBD

SUMMARY:
Interventional study using Cannabidiol containing cigarettes as replacement of usual cigarettes

Reduction of enforcement measures, improved acute treatment, harm reduction, and improvement of psychotic symptoms

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia or Related Disorders
* PANNS > 21,
* Tobacco-smokers
* inpatient status
* within age 18 - 65 years
* German-speaking

Exclusion Criteria:

* personality disorder
* non-smokers
* organic psychotic diseases
* breast feeding
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in psychotic symptoms | 1 Months (acute therapy), 6 Months (Follow up)
  To measure changes in psychotic symptoms weekly PANNS (Positive and Negative Syndrome Scales) are used. This is a validated medical scale used for measuring symptom severity of patients with schizophrenia. The patient is rated from 1 to 7 on 30 different symptoms based on a clinical interview. Minimum Score = 30, Maximum Score = 210 Points. Lower Scores mean less positive / less negative / less general psychopathological symptoms, which is better. Higher scores mean more postive / negativ / general psychopathological symptoms.
Change in violent behaviour. | 1 Month (acute therapy), 6 Months (Follow up)
  Violent behaviour will be assessed through clinical staff via the The Brøset Violence Checklist. It is a clinical evaluation indicating the presence or absence of violent behaviour. The scale consists of 6 items. Minimum score = 0, Maximum score = 6. The lower the score, the better. A low score indicates a lower potential of violent behaviour and lower actual violent behaviour.
Change in depressive Symptoms | 1 Month (acute therapy), 6 Months (Follow up)
  To measure changes in depressive Symptoms weekly BDI-II (Becks Depression Inventory) will be conducted (minimum = 0 points, maximum = 63 points). A higher score means more severe depression.
Change in subjective well being under neuroleptic medication | 1 Month (acute therapy), 6 Months (Follow up)
  Subjective Well-Being under Neuroleptics Scale short form (SWN-K) will be used to assess individual well-being on a weekly basis. (Minimum = 20, Maximum = 120 points). Higher scores mean higher subjective well-being.
Change of necessary neuroleptic medication | 1 Month (acute therapy), 6 Months (Follow up)
  We will register the patients neuroleptic medication. For the conversion of the participants' antipsychotic medication the Defined Daily Dose method by Leucht et al. (2016) was applied. Each participants' antipsychotic medication was converted to olanzapine equivalents in mg per day using the antipsychotic dose conversion calculator provided by Leucht and colleagues (Leucht et al., 2020).

SECONDARY OUTCOMES:
Total number of Isolation-Events (enforcement measures) | 1 Month (acute therapy), 6 Months (Follow up)
  The total number of necessary Isolations of participants in CBD-arm and non-CBD-arm will be compared. The total number of actual isolation events will be compared
Total number of enforced medication-events (enforcement measures) | 1 Month (acute therapy), 6 Months (Follow up)
  The number of necessary events of enforced medication of participants in CBD-arm and non-CBD-arm will be compared. The total number of actual enforced medication-events will be compared.
Tobacco use | 1 Month (acute therapy), 6 Months (Follow up)
  Number of normal tobacco cigarettes and CBD-Cigarettes will be measured by a daily self-reporting-scale of the participants.
Cannabis use | 1 Month (acute therapy), 6 Months (Follow up)
  Number of cannabis-joints will be measured by weekly self-reports of the participants.
Correlation of CBD and THC levels with psychotic symptoms via PANSS | 1 Month (acute therapy), 6 Months (Follow up)
  The study aims to correlate CBD and THC whole blood levels with psychotic symptoms via PANSS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Undine Lang, Prof. Dr., Principal Investigator — Director
Locations (1):
- Universitäre Psychiatrische Kliniken, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kock P, Lang E, Trulley VN, Dechent F, Mercer-Chalmers-Bender K, Frei P, Huber C, Borgwardt S. Cannabidiol Cigarettes as Adjunctive Treatment for Psychotic Disorders - A Randomized, Open-Label Pilot-Study. Front Psychiatry. 2021 Nov 4;12:736822. doi: 10.3389/fpsyt.2021.736822. eCollection 2021. PMID 34803760